CLINICAL TRIAL: NCT04262375
Title: A Phase 2 Study of Durvalumab (MEDI4736) and Oleclumab (MEDI9447) in Multi-Cancer Populations With Correlation to Clinical, Molecular and Immunologic Parameters With DNA MethylaTION (DOMINATION)
Brief Title: A Phase 2 Study of Durvalumab (MEDI4736) and Oleclumab (MEDI9447) in Multi-Cancer Populations With Correlation to Clinical, Molecular and Immunologic Parameters With DNA MethylaTION
Acronym: DOMINATION
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Overall clinical activity (ORR) for oleclumab + durvalumab is minimal across tumor types and does not support further evaluation of this doublet.
Sponsor: University Health Network, Toronto (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOMINATION; 19-6281 (Other: University Health Network)
Record Dates: First submitted 2020-02-05; First posted 2020-02-10 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Non Small Cell Lung Cancer; Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab and Oleclumab (Experimental): A single dose level for oleclumab and durvalumab will be used, comprising of Oleclumab 3000 mg IV Q2W for 4 doses, then Q4W AND Durvalumab 1500 mg IV Q4W
  Interventions: Biological: Durvalumab; Biological: Oleclumab

INTERVENTIONS:
Biological: Durvalumab — Durvalumab is a human immunoglobulin G (IgG)1 kappa monoclonal antibody directed against human PD-L1. Durvalumab selectively binds human PD-L1 with high affinity and blocks its ability to bind to PD-1 and cluster of differentiation (CD)80. The fragment crystallizable (Fc) domain of durvalumab contains a triple mutation in the constant domain of the IgG1 heavy chain that reduces binding to the complement component C1q and the Fc gamma receptors responsible for mediating antibody dependent cell mediated cytotoxicity.
  Other Names: IMFINZI
Biological: Oleclumab — Oleclumab is a human immunoglobulin G1 lambda monoclonal antibody (mAb) with a triple mutation in the heavy chain constant region for reduced effector function. Oleclumab selectively binds to cluster of differentiation 73 (ecto-5'-nucleotidase) (CD73) and inhibits CD73-associated ectonucleotidase activity, thereby inhibiting the CD73-mediated production of immunosuppressive adenosine. Extracellular adenosine contributes to the immunosuppressive effects of both regulatory T cells and myeloid derived suppressor cells, among others. This, in turn, leads to increased antitumor immunity.

SUMMARY:
This is a Phase II, prospective, non-randomized, open-label trial involving cancer patients with known inflamed tumor types. Patients with previously treated advanced/metastatic non-small cell lung cancer or renal cell cancer will be recruited in near equal distribution. All patients must have documented response or prolonged stable disease to previous immunotherapy. At present, we plan to enrol 55 patients, to be treated with durvalumab and oleclumab. The regimen will consist of durvalumab 1500 mg given by vein every 4 weeks and oleclumab 3000 mg given by vein every 2 weeks x 4 doses then IV every 4 weeks till disease progression, withdrawal of subject consent, or another reason for discontinuation. Estimated total duration from time to first subjects consent to last subject's last visit is approximately 36 months.

DETAILED DESCRIPTION:
Study Hypotheses:

1. Circulating free methylated DNA immunoprecipitation and high-throughput sequencing (cfMeDIP-seq) can yield cancer type-agnostic predictive biomarker(s) of response and/or toxicity in subjects receiving this combination.
2. The combination of oleclumab (anti-cluster of differentiation [CD]73 monoclonal antibody) with durvalumab (anti programmed cell death ligand 1 [PD-L1]) will demonstrate adequate safety, tolerability, and antitumor activity in subjects with metastatic non-small-cell lung cancer (NSCLC) and renal cell cancer (RCC) previously treated with checkpoint inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of screening or age of consent according to law
2. Life expectancy of at least 12 weeks
3. Written informed consent and any locally required authorization obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
4. ECOG 0 or 1
5. Weight ≥35kg
6. Subjects diagnosed with histologically or cytologically confirmed non small cell lung (NSCLC) or renal cell carcinoma (RCC)
7. Subjects must have at least 1 measurable lesion according to RECIST version 1.1.
8. Archival tumor formalin-fixed, paraffin-embedded (FFPE) specimens for correlative biomarker studies are required (1 H&E and 15 unstained slides). Subjects with insufficient archived tumor samples are still eligible, pending discussion with the principal investigator on a case by case basis
9. Adequate organ and marrow function
10. Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception from screening to 90 days after the final dose of study treatment
11. Nonsterilized male subjects who are sexually active with a female partner of childbearing potential must use a male condom with spermicide from screening to 90 days after receipt of the final dose of study treatment

Exclusion Criteria:

1. Receipt of any conventional or investigational anticancer therapy within 21 days or palliative radiotherapy within 14 days prior to the scheduled first dose of study treatment
2. Prior receipt of any agents targeting CD73, including patients treated with adenosine receptor antagonists, CD39 or CD73 inhibitors
3. Prior receipt of any innate immune agonists
4. Patients with NSCLC with known activating EGFR mutations or ALK translocations
5. Concurrent enrollment in another therapeutic clinical study. Enrollment in observational studies will be allowed
6. Any toxicity (excluding alopecia) from prior standard therapy that has not been completely resolved to baseline at the time of consent
7. Subjects with a history of Grade 3 or greater thromboembolic events in the prior 12 months or thromboembolic event of any grade with ongoing symptoms
8. Subjects with prior history of myocardial infarction, transient ischemic attack, congestive heart failure ≥ Class 3 based on New York Heart Association Functional Classification or stroke within the past 3 months prior to the scheduled first dose of study treatment
9. Active or prior documented autoimmune disorders within the past 3 years prior to the scheduled first dose of study treatment
10. HIV, Hep A, B, or C
11. History of primary immunodeficiency, solid organ transplantation, or active tuberculosis
12. Known allergy or hypersensitivity to investigational product formulations
13. History of more than one event of infusion related reactions (IRR) requiring permanent discontinuation of IV drug treatment
14. Active grade 3 or greater edema
15. History of Grade 3 or greater thromboembolic events in the prior 12 months or thromboembolic event of any grade with ongoing symptoms
16. Uncontrolled intercurrent
17. Any history of untreated leptomeningeal disease or cord compression
18. Untreated CNS metastatic disease
19. Current or prior use of immunosuppressive medication within 14 days prior to the scheduled first dose of study treatment
20. Receipt of live, attenuated vaccine within 30 days prior to the scheduled first dose of study treatment
21. Major surgery within 28 days prior to scheduled first dose of study treatment or still recovering from prior surgery
22. Females who are pregnant, lactating, or intend to become pregnant during their participation in the study
23. Subjects who are involuntarily incarcerated or are unable to willingly provide consent or are unable to comply with the protocol procedures
24. Any condition that would interfere with the evaluation of the study regimen or interpretation of patient safety or study results
25. Any condition that would interfere with safe administration or evaluation of the investigational products or interpretation of subject safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Association between cfMeDIP and Response (defined as either complete response, partial response, or stable disease ≥ 4 cycles, as per RECIST 1.1. Association between cfMeDIP and Toxicity (defined as ≥ Grade 2 immune- adverse event (AE) as per CTCAE 5.0). | 3 years
  To identify cfMeDIP-seq-based predictive signature(s) that are correlated with specific outcome to durvalumab and oleclumab such as response/resistance or occurrence of toxicity in non-small cell lung cancer (NSCLC) and renal cell carcinoma (RCC)
Objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | 3 years
Disease control rate (DCR) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | 3 years
Duration of response (DoR) | 3 years

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs) | 3 years
  To assess the safety and tolerability of durvalumab and oleclumab in specific disease states in NSCLC and RCC
Overall survival (OS) or progression-free survival (PFS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Albiruni Razak, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No